CLINICAL TRIAL: NCT04929587
Title: Analysis of Influencing Factors of Preoperative Frailty in Elderly Patients With Gastric Cancer Based on the Health Ecology Theory
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lingyu Ding, Clinical nurse, Nanjing Medical University
Other Study IDs: LDing
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer; Frailty
MeSH Terms: conditions — Stomach Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a observational research, there is no intervention — This is a observational research, there is no intervention

SUMMARY:
Frailty is common in patients with gastric cancer undergoing surgical treatment. Preoperative frailty can lead to many adverse outcomes in patients after surgery. This study aims to comprehensively and systematically analyze the influencing factors of preoperative frailty in patients with gastric cancer based on the health ecology theory , to change some critical variable factors in the future, improving the overall prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer
* Age over 60 years old
* With clear surgical indication

Exclusion Criteria:

* Malignant tumors in other parts of the body
* Severe cardiopulmonary complications
* Receive palliative surgery
* Have received preoperative radiotherapy and chemotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged over 60 years old and who have gastric cancer with clear surgical indications
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Frailty assessed by Frailty Phenotype (FP) | preoperative period
  The total score is 0~5, and a score of 0~3 is considered as frailty.

SECONDARY OUTCOMES:
Nutrition assessed by Nutrition Risk Screening 2002 (NRS2002) | preoperative period
  NRS2002 comprises 3 components: nutritional status, disease status and age, with a total score ranging from 0 to 7. A score of ≥3 is considered to be at nutritional risk.
Anxiety and depression assessed by Hospital Anxiety Depression Scale (HADS) | preoperative period
  HADS contains 2 subscales: anxiety and depression subscales. Each subscale consists of 7 items, with a total score ranging from 0 to 21. A score of each subacale reaches 8 or more is regarded as the presence of anxiety or depression.
Social support assessed by Social Support Rate Scale (SSRS) | preoperative period
  SSRS contains 10 items and 3 dimensions, which are objective support, subjective support, and support utilization, with higher scores indicating higher degrees of the corresponding dimensions.
Familial caring degree assessed by Family Concern Index Questionnaire (APGAR) | preoperative period
  The total score ranges from 0 to 10, and a score of ≤6 is considered as having family dysfunction.
Sleep assessed by Pittsburgh Sleep Quality Index (PSQI) | preoperative period
  A total score range from 0 to 21, a score of 0~5 indicates "very good" sleep quality; a score of 6~10 indicates "good" sleep quality; a score of 11~15 indicates "poor" sleep quality; a score of 16~21 indicates "very poor" sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided